CLINICAL TRIAL: NCT04733313
Title: Comparison of Ultrasound Guided Quadratus Lumborum Block-2 and Quadratus Lumborum Block-3 for Postoperative Pain in Cesarean Section
Brief Title: Effect of Quadratus Lumborum Block in C/S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ferit Yetik, medical doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-7/8
Record Dates: First submitted 2021-01-24; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Cesarean Section Complications; Block; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quadratus lumborum-2 (Active Comparator)
  Interventions: Procedure: ultrasound guıded quadratus lumborum block
- quadratus lumborum-3 (Active Comparator)
  Interventions: Procedure: ultrasound guıded quadratus lumborum block

INTERVENTIONS:
Procedure: ultrasound guıded quadratus lumborum block — Administering local aneshtetic agent with a block needle using the in-plane technique, bilaterally. Lumbar interfascial triangle, where the middle lumbar fascia joins the deep lamina of the posterior layer on the lateral border of the erector spinae was targeted as the optimal point of injection.

SUMMARY:
to compare postoperative analgesic effects of USG guided QLB-2 and QLB-3 blocks after C/S. We hypothesized that QLB-3 may be more effective for pain relieving than QLB-2 after C/S.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy with a gestation of 37-41 weeks parturients who were scheduled for elective cesarean delivery under general anesthesia
* obtained patients informed consent

Exclusion Criteria:

* inability to comprehend
* bleeding diathesis
* allergy to the study agents
* localized infection
* block failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Assesment of postoperative pain | during 24 hour after surgery
  measure of the visual analog scale at rest and dynamic after surgery

SECONDARY OUTCOMES:
need of analgesic | during 24 hour after surgery
  total number of PCA demands

CONTACTS AND LOCATIONS:
Locations (1):
- Healt Science University Bursa Training and Research Hospita, Bursa, Yildirim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No